CLINICAL TRIAL: NCT01094665
Title: Phase 1 Study of MRI Targeted Focal Laser Thermal Therapy of Prostate Cancer
Brief Title: MRI Targeted Focal Laser Thermal Therapy of Prostate Cancer
Acronym: FLTT002
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0689-C
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focal Laser Thermal Therapy (Experimental): Thermal therapy delivered to lesion visible on MRI.
  Interventions: Procedure: MRI Targeted Focal Laser Thermal Therapy

INTERVENTIONS:
Procedure: MRI Targeted Focal Laser Thermal Therapy — A 980nm wavelength diode laser will be fired for up to 30 minutes. Temperature probes will be inserted to ensure that the local temperature does not exceed 55 degrees Celsius for more than 5 minutes.

SUMMARY:
The primary objective of this study is to evaluate the safety and feasibility of Magnetic Resonance Image (MRI) guided focal prostate cancer laser thermal ablation in males, ages 40-80 with biopsy confirmed early clinical stage prostate cancer (T1c or T2a) with an identifiable lesion on mutliparametric MRI, with a Prostate Specific Antigen (PSA) of < 15ng/ml, who have not yet undergone pelvic radiation or hormonal deprivation therapy.

DETAILED DESCRIPTION:
This is a single center, single arm, open-label study to evaluate the safety and feasibility of MRI guided focal prostate cancer laser ablation in patients with a focus of prostate cancer who has not yet received treatment for their cancer. Patients fulfilling the inclusion criteria and having none of the clinical exclusion criteria will be enrolled into the study after they (or their legal representative) have signed the informed consent form. No control group will be utilized and all patients will receive MRI guided FLA for their focal prostate cancer. As part of the screening process, patients will provide a medical history and undergo a physical examination, including a digital rectal examination (DRE). At the first visit, patients will also be given a copy of the informed consent, and a copy of quality of life and performance questionnaires to assess urinary, rectal, and erectile functions (IPSS questionnaire for urinary, IIEF5 questionnaire for erectile function, for all). MR imaging at visit 2 will serve to determine if a single site of prostate cancer can be localized. At visit 3, 12 cores transrectal us guided prostate biopsy will confirm yet again that this is a unilateral, unifocal histologically proven tumour in the site recognized on the MRI. On preoperative examination (visit 4) - blood and urine samples will be taken prior to procedure. Visit 5 - the focal treatment will be performed under regional or general anesthesia, or conscious sedation, (as determined by the anesthesiologist) in the TGH research 1.5T MRI suite. MR guided FLA procedure is similar to MR guided brachytherapy, with fibers and probes inserted transperineally outside the bore of the MR and then the patient is moved inside the bore to verify position before deploying the laser. The treatment is expected to last 2-3 hours, and patients expected to have no pain during the whole procedure. Laser ablation will be monitored using MR thermometry14, 15.An MRI scan will be done immediately after the ablation, as initial assessment for ensuring complete treatment of the target volume, as well as ensuring that treatment does not extend to critical structures.

The size and location of the lesion will be compared to the planned target volume and the proximity of the lesion to the urethra and rectum. If the lesion does not encompass the target volume, and is still a safe distance from either critical structure, FLA may be continued.

On day 3, 7, 30, and 120 following the procedure, patients will be assessed for clinical signs of urinary, rectal, and erectile complications and will complete validated self-assessment tools on these functions. Free/Total PSA will be monitor on visit -1 and after the treatment on day 7, 30 and 120, in order to try to understand the effect of FLA on PSA. Four months after the focal procedure, a further 12 cores biopsy, plus 2 cores aimed to the ablated lesion will then be preformed to verify the oncological effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men 45-80 years of age;
* Histologically proven prostate carcinoma;
* Prostate cancer clinical stage T1c and T2a
* Prostate MRI must confirm area suspicious for cancer in the sector of the positive biopsy;
* Prostate specific antigen (PSA) level less than 15 ng/mL
* 12 cores biopsy, with histologically proven prostate carcinoma, in the suspicious region on MRI.
* IPSS and IIEF complete prior to procedure
* Life expectancy of greater than 5 years, based on co-morbidity not related to prostate cancer.

Exclusion Criteria:

* Medically unfit for focal therapy of the prostate
* Patients who are unwilling or unable to give informed consent;
* Patients who have received androgen suppression therapy
* Patients who have received or are receiving chemotherapy for prostate carcinoma;
* Patients previously treated with surgery to the prostate (traditional, endoscopic or minimally invasive including HIFU, TUNA, RITA, microwave, TURP, cryotherapy or any curative treatment
* Patients who have undergone radiation therapy for prostate cancer or to the pelvis
* Any condition, or history of illness or surgery that, in the opinion of the Investigator, might confound the results of the study or pose additional risks to the patient (e.g. significant cardiovascular conditions or allergies);
* Patients with a history of non compliance with medical therapy and/or medical recommendations;
* Patients who are unwilling or unable to complete the patient self-assessment questionnaires;
* Chronic or acute prostatitis, neurogenic bladder, urinary tract infection, sphincter abnormalities, or any other symptom that prevents normal micturition.
* Patients who have participated in a clinical study and/or received treatment with an investigational treatment and/or product within the past 90 days;
* If the patient is unable to undergo regional anesthesia
* Patients with contraindication to MRI (i.e. pacemaker, hip prosthesis, severe claustrophobia, brain aneurysm clip, allergy to MRI contrast agent)
* Any condition, or history of illness that, in the opinion of the investigator will confound or increase the patient risk during the study

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-11; Primary Completion 2015-10-08 (Actual); Study Completion 2015-10-08 (Actual)

PRIMARY OUTCOMES:
Transrectal Ultrasound Guided Prostate Biopsy | 4 Months Post Treatment
  A 12 core biopsy, plus 2 cores aimed at the ablated lesion will then be preformed to verify the oncological effectiveness of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, University Health Network, Toronto, Ontario, Canada